CLINICAL TRIAL: NCT01777971
Title: The Effect of a Large-volume Paracentesis on Fatigue, Sleep, and Quality of Life in Cirrhosis
Status: Withdrawn | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: R11-00672
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Cirrhosis; Hepatic Encephalopathy; Ascites; Fatigue
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Ascites; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with cirrhosis: Male and female subjects who have cirrhosis of the liver and diuretic-resistant ascites (based on International Ascites Clib criteria) and have been evaluated and approved to have a large-volume paracentesis as part of standard of care treatment.

SUMMARY:
Ascites is the accumulation of fluid within the peritoneal cavity of the abdomen. It is a frequent complication of cirrhosis that is associated with significant morbidity and poor quality of life. Large-volume ascites has been associated with impaired pulmonary function. In a previous study, the presence and severity of ascites were determined to be significant determinants of fatigue.

In this study, we will determine whether large-volume ascites contributes to fatigue by assessing the response to drainage of ascites by means of a procedure called large-volume paracentesis. We hypothesize that treatment of ascites with a single large-volume paracentesis leads to decreased fatigue and improved quality of life and that this improvement is associated with improved sleep pattern.

20 patients with cirrhosis with refractory ascites requiring regular drainage of ascites fluid by large-volume paracenteses will be recruited for the study. All patients will undergo a complete clinical and physical examination for liver function, including blood tests. Hepatic encephalopathy, a change in mental status associated with liver dysfunction, will be assessed by obtaining historical data and by means of simple bedside neuropsychological examinations.

Study visits will take place on two consecutive days, with each visit lasting approximately 2-3 hours. Immediately prior to a large-volume paracentesis, patients will complete standardized questionnaires for fatigue severity, quality of life, quality of sleep, and a physical assessment of fatigue by means of a 6-minute walk test. Repeat evaluations will be performed 1 day after the procedure. Statistical analysis will then be performed to determine the effect of the paracentesis on the various clinical assessments.

DETAILED DESCRIPTION:
The study design is a prospective observational analysis. Subjects who have been deemed candidates for a large-volume paracentesis, based on clinical criteria and who meet the above-referenced inclusion and exclusion criteria will be recruited to participate in this study. Study visits will take place on 2 consecutive days. Each study visit will last approximately 2 to 3 hours. The first assessment day will occur immediately prior to an electively-scheduled large-volume paracentesis. The second assessment will occur one day later.

Once enrolled, all subjects will undergo a baseline assessment of liver function. Medical records will be reviewed to determine etiology of cirrhosis, history of variceal bleeding, history of spontaneous bacterial peritonitis, history of hospitalization for hepatic encephalopathy, and use of and clinical response to treatment with lactulose, neomycin, and/or rifaximin. Body mass index and grade of ascites (grade 1, mild ascites; grade 2, moderate ascites; grade 3, massive or tense ascites) will be determined based on physical examination. History or presence of asterixis will be recorded. Severity of hepatic encephalopathy will be graded according to the West-Haven criteria and further assessed by neuropsychological testing (discussed in further detail below). Baseline serum laboratory analyses will be obtained, including the following: aspartate aminotransferase, alanine aminotransferase, total bilirubin, albumin, blood urea nitrogen, creatinine, prothrombin time and international normalized ratio, and platelet count. Based on these serum studies, the Child-Pugh score and Model for End-Stage Liver Disease score will be calculated.

After baseline assessments are obtained, the six-minute walk test and a series of questionnaires (discussed in further detail below) to assess fatigue, sleep, and quality of life will be performed on study day 1, immediately prior to the paracentesis, and then repeated one day after the paracentesis. Note that neither the six-minute walk test nor the neuropsychological testing or questionnaires are considered standard of care for patients requiring large-volume paracentesis and these will be performed exclusively for research purposes.

ELIGIBILITY:
Inclusion Criteria:

Subjects with cirrhosis (based on clinical, laboratory, radiologic evaluation, and liver biopsy, when available) with diuretic-resistant refractory ascites, based on International Ascites Club criteria.[2,31] Specific criteria used for inclusion will be subjects with ascites that cannot be stabilized despite intensive diuretic therapy (e.g., 400 mg of spironolactone with 160 mg of furosemide per day) and dietary sodium restriction (90 mmol of sodium per day) with reappearance of grade 2 or 3 ascites within 4 weeks of mobilization (defined as decrease of ascites at least to grade 1). All subjects must provide separate written consent to undergo a large-volume paracentesis.

Exclusion Criteria:

Subjects will not be eligible for the study if they: (1) have been hospitalized in the previous 1 month for gastrointestinal bleeding, infection, or renal failure; (2) are unable to independently ambulate or have had unstable angina or myocardial infarction within the previous 1 month, as these are contraindications to participating in the 6-minute walk test; (3) are unable to participate in neuropsychological tests or questionnaires; (4) are receiving interferon therapy; (5) have a history of alcohol abuse within the previous 6 months; (6) have a diagnosis of a primary neurologic disorder or uncontrolled psychiatric disorder; or (7) are receiving psychotropic medications such as benzodiazepines and anti-epileptic drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis with diuretic-resistant refractory ascites (based on International Ascites Club criteria)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Fatigue | 10 min
  Patients undergo 6-minute walk test and fill out Fisk Impact Scale (Fatigue Questionnaire)

SECONDARY OUTCOMES:
Hepatic Encephalopathy | 10 min
  Patients undergo psychometric testing that involves Trail Making Test and Digit Symbol Substitution Test.
Quality of Life | 5 min
  Patients fill out Medical Outcomes Study Short Form 36 questionnaire
Daytime Sleepiness | 5 min
  Patients fill out Epworth Sleepiness Scale questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States